CLINICAL TRIAL: NCT01924845
Title: A Phase 3 Switchover Study of the Efficacy and Safety of BMN 701 (GILT-tagged Recombinant Human GAA) and Long-Term Study for Extended Treatment in rhGAA Exposed Subjects With Late-onset Pompe Disease
Brief Title: BMN 701 Phase 3 in rhGAA Exposed Subjects With Late Onset Pompe Disease (INSPIRE Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 701-301; 2013-001768-48 (EudraCT Number)
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Late-onset Pompe Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMN 701 20 mg/kg (Experimental): BMN 701 IV Infusion 20mg/kg every 2 weeks for 24 weeks followed by an optional extension of 240 weeks (total duration of therapy 264 weeks)
  Interventions: Drug: BMN 701

INTERVENTIONS:
Drug: BMN 701 — BMN 701 20 mg/kg for intravenous administration over approximately 4 hours every 2 weeks over a 24-week Treatment Period (total of 13 doses), and every 2 weeks over a 240-week Extension Period (up to 120 additional doses).

SUMMARY:
Study 701-301 is a single-arm, open-label, switchover study in patients with late-onset Pompe disease who have been receiving treatment with recombinant human acid alpha-glucosidase (rhGAA) for 48 weeks or longer. Ambulatory patients who have mild to moderate respiratory impairment will switch directly to receive BMN 701 20 mg/kg by IV infusion every other week. All participants will receive active drug. No dose of existing therapy will be missed - experimental drug is started immediately.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent, after the nature of the study has been explained, and prior to any study-related procedures.
* Diagnosed with late-onset Pompe disease based on 2 currently or previously documented GAA gene mutations, and endogenous GAA activity <75% of the lower limit of the normal adult range reported by the testing laboratory, as assessed by dried blood spot or whole blood assay.
* Has received prior treatment with commercial rhGAA as defined by ALL of the following:

  1. has received treatment with commercial rhGAA for ≥ 48 weeks (but no more than 20% of the study population can have received treatment for ≥ 6 years).
  2. has received > 80% of all scheduled treatments in the prior 48 weeks and ≥ 4 out of the prior 6 scheduled treatments.
  3. has received and completed the last two infusions without a drug-related adverse event resulting in dose interruption.
  4. has received last treatment of commercial rhGAA ≥ 10 and ≤ 31 days prior to anticipated initiation of treatment with BMN 701.
* ≥ 18 years of age at the time of enrollment in the study.
* Sexually active subjects must be willing to use two known effective methods of contraception while participating in the study and for at least 4 months following the last dose of BMN 701.
* Females of childbearing potential must have a negative pregnancy test at Screening and Baseline visits and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
* Has ≥ 30% predicted upright FVC and < 80% predicted upright FVC.
* Has ≤60% predicted MIP.
* Is able to ambulate ≥75 meters and ≤500 meters on the 6MWT conducted during the Screening visit (use of assistive devices such as walker, cane, or crutches, is permitted with consistent use throughout the study).
* Is willing and able to comply with all study procedures.

Exclusion Criteria:

* Use of any investigational product or investigational medical device within 4 weeks prior to Screening, or requirement for any investigational agent other than BMN 701 prior to completion of at least the first 24 weeks of all scheduled study assessments.
* Received any investigational medication for Pompe disease within the prior 12 months.
* Has a diagnosis of diabetes and/or is currently being treated with or anticipated to require treatment with hypoglycemic agents during the course of the study.
* Has been treated with any immunosuppressive medication other than glucocorticosteroids within the prior 12 months.
* Requires noninvasive ventilatory support while awake and in the upright position.
* Has previously been enrolled to this study.
* Breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Concurrent disease, medical condition, or extenuating circumstance that, in the opinion of the Investigator, might compromise subject safety, study treatment compliance and completion of the study, or the integrity of the data collected for the study.
* Has known hypersensitivity to BMN 701 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Monitor, Study Director — BioMarin Pharmaceutical
Locations (22):
- United States (8):
  - Neuromuscular Research Centre, Phoenix, Arizona
  - University of California, Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
- Antwerp University Hospital (UZA), Edegem, Belgium
- France (2):
  - Hôpital Raymond Poincaré, Garches
  - CHU de la Timone, Marseille
- Germany (3):
  - Villa Metabolica, ZKJM MC University Mainz, Mainz
  - Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster
- Italy (2):
  - Azienda Ospedaliera Universitaria Policlinico "G. Martino" - Messina, Messina, ME
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
- Erasmus MC University Medical Center, Rotterdam, Netherlands
- Centro Hospitalar de Sao Joao, EPE, Porto, Portugal
- United Kingdom (4):
  - University Hospital Birmingham, Birmingham
  - Royal Free Hospital, London
  - National Hospital for Neurology and Neurosurgery, London
  - Salford Royal NHS Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 31-day Screening and Baseline Period (26-day Screening Period, a 5-day Baseline/Enrollment Period), a 24-week Treatment Period, and a 30-day Safety Follow-up Period. Following the Screening and Baseline assessments, qualified subjects were enrolled in the study.
Groups:
- BMN 701 20 mg/kg: BMN 701 20 mg/kg
Period: Overall Study
Arm/Group | BMN 701 20 mg/kg
Started | 24
Completed | 18
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | BMN 701 20 mg/kg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (13.27)
Age, Customized [Count of Participants; unit: Participants]
  18-65 | 22
  > 65 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1
  Germany | 9
  United Kingdom | 7
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted Maximum Inspiratory Pressure (MIP)
Description: Pulmonary function test: Percent Predicted Maximum Inspiratory Pressure
Time Frame: Baseline, Week 24
Population: Full Analysis Set. Please note the Overall Number of Participants reflects the number of patients in the Analysis Population, while the Number Analyzed of patients at specific visit in the Outcome Measure Table reflects the participants who had data at that visit .
Measure: Mean (Standard Deviation); unit: Percent Predicted
Groups:
- BMN701 20 mg/kg: BMN701 20 mg/kg
Arm/Group | BMN701 20 mg/kg
Number analyzed (Participants) | 18
Percent Predicted
  Baseline | 50.0 (17.5)
  Change from Baseline to Week 24 | 2.2 (8.3)

2. Secondary Outcome: Percent Predicted Maximum Expiratory Pressure (MEP)
Description: Pulmonary function test: Percent Predicted Maximum Expiratory Pressure
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | BMN701 20 mg/kg
Number analyzed (Participants) | 18
Percent Predicted
  Baseline | 38.9 (12.3)
  Change from Baseline to Week 24 | 3.1 (8.7)

3. Secondary Outcome: 6 Minute Walk Test (Meters)
Description: Distance walked within 6 minutes
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | BMN701 20 mg/kg
Number analyzed (Participants) | 17
Meter
  Baseline | 345.8 (95.3)
  Change from Baseline to Week 24 | 26.1 (40.6)

4. Secondary Outcome: Percent Predicted Upright Forced Vital Capacity (FVC)
Description: Pulmonary function test: Percent Predicted Upright Forced Vital Capacity
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | BMN701 20 mg/kg
Number analyzed (Participants) | 18
Percent Predicted
  Baseline | 60.7 (15.1)
  Change from Baseline to Week 24 | -3.7 (4.4)

5. Secondary Outcome: Number of Participants With Non-Serious AEs
Description: Number of participants with non-serious Adverse Events. Data is taken at final time point of Week 24, compared to baseline. For full AE data, please see AE section.
Time Frame: Baseline through Week 24 +4 weeks follow-up
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN701 20 mg/kg
Number analyzed (Participants) | 24
Participants | 23

ADVERSE EVENTS:
Time Frame: 28 weeks (24 weeks trial + 4 weeks follow up)
Arm/Group | BMN 701 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 10/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 20 mg/kg (N=24)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 20 mg/kg (N=24)
Palpitations (Cardiac disorders) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 8 (22)
Vomiting (Gastrointestinal disorders) | 4 (7)
Chest discomfort (General disorders) | 2 (3)
Chills (General disorders) | 4 (6)
Fatigue (General disorders) | 5 (8)
Pain (General disorders) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (5)
Pharyngitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 5 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 16 (165)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Dizziness (Nervous system disorders) | 8 (12)
Headache (Nervous system disorders) | 13 (50)
Lethargy (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cold sweat (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Complete efficacy analyses were not able to be completed due to early study termination; however, efficacy results from interim analysis at week 24 are available, and thus have been reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes